CLINICAL TRIAL: NCT01748786
Title: Emotional Resilience in Fibromyalgia: A Pilot Study of Web-based Treatment
Brief Title: Online Mindfulness Training Versus Health Education for Fibromyalgia
Acronym: EGIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Arizona Institute for Mental Health Research (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZIMHR-01
Record Dates: First submitted 2012-12-07; First posted 2012-12-13 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Mindfulness; On-line intervention; Chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Emotion Regulation (Experimental): 12 on-line modules targeting social and emotional regulation through mindfulness training
  Interventions: Behavioral: Mindfulness Emotion Regulation
- Placebo (Placebo Comparator): 12 on-line modules providing information regarding health behaviors
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Mindfulness Emotion Regulation — 12 on-line modules provide didactic information and practice instructions re: mindfulness meditation for pain and distress
  Arms: Mindfulness Emotion Regulation
Other: Health Education — 12 on-line modules that provide information regarding health behaviors, but no information regarding how to put behaviors into practice
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare an online 12-module intervention designed to improve emotion regulation and social relations via mindfulness training with a 12-module program that provides information about health behaviors to individuals with fibromyalgia. The mindfulness training program is expected to produce greater day-to-day improvements than the education condition in individuals' efficacy for coping with pain and stress, positive and negative affect, and positive engagement in social relations assessed via online diaries completed each evening during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Self-report of physician diagnosis of fibromyalgia
* Able to read and understand English
* Daily access to the internet

Exclusion Criteria:

* Self-report of more than 5 past episodes of depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Daily Positive affect (10 items rated 1-5, averaged) and negative affect (10 items rated 1-5, averaged) | Daily during 6-week intervention
  Trajectory of change in positive affect over the course of the trial is assessed via daily diaries. Positive and negative affect subscales are assessed daily with the Positive (10 items) and Negative (10 items) Affect Schedule (PANAS; Watson, Clark, & Tellegen, 1988).
Daily Pain Coping Efficacy (1 item rated 1-5) and Stress Coping Efficacy (2 item rated 1-5, averaged) | Daily over 6-week intervention
  Trajectory of change over the course of the intervention via daily diary reports. Pain and stress coping efficacy (PCE and SCE) are assessed with 2 items each, with items combined to form a mean score for PCE and for SCE (Johnson, Zautra, & Davis 2006). "The first was "How satisfied are you with how you coped with your symptoms (stress)?" referring to that day, rated on a 5-point Likert scale ranging from 1=very dissatisfied to 5=very satisfied. The second item was "If you had this level of pain (stress) again, how certain are you that you would be able to cope well with its negative aspects?" rated on a 5-point Likert scale, ranging from 1=very uncertain to 5 = very certain.

SECONDARY OUTCOMES:
Daily Enjoyment (1 item rated 1-5) and Stressfulness (1 item rated 1-5) of Family Relations | Daily during 6-week intervention
  Trajectory of change over the course of the trial via daily diaries. Daily family relations were assessed by two items asking how enjoyable (1 item) and how stressful (1 item) individuals found the time they spent with family on that day, with each item rated on a 4-point scale ranging from 1=not at all to 4 = extremely. These items were drawn from the Inventory of Small Life Events scale (Zautra, Guarnaccia, & Dohrenwend, 1986)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

REFERENCES:
- [Derived] Davis MC, Zautra AJ. An online mindfulness intervention targeting socioemotional regulation in fibromyalgia: results of a randomized controlled trial. Ann Behav Med. 2013 Dec;46(3):273-84. doi: 10.1007/s12160-013-9513-7. PMID 23670111